CLINICAL TRIAL: NCT07371780
Title: Heart Failure Center Accreditation Program (HF-CAP) in China: A Prospective Multicenter Cluster Randomized Controlled Trial
Brief Title: Heart Failure Center Accreditation in China (HF-CAP Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B2025 -675
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-CAP Intervention (Experimental): Hospitals assigned to this arm will implement the Heart Failure Center Accreditation Program (HF-CAP).
  The intervention includes standardized heart failure care processes, multidisciplinary team-based management, regular training of healthcare professionals, patient and caregiver education, structured discharge planning, and post-discharge follow-up, as well as continuous quality monitoring and feedback. Patients hospitalized for heart failure in these hospitals will receive care under the HF-CAP framework.
  Interventions: Other: Heart Failure Center Accreditation Program (HF-CAP)
- Usual Care (Active Comparator): Hospitals assigned to this arm will provide usual care for patients hospitalized with heart failure.
  Usual care is delivered according to local clinical practice and existing guidelines, without implementation of the Heart Failure Center Accreditation Program (HF-CAP) or additional quality improvement interventions.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Heart Failure Center Accreditation Program (HF-CAP) — The Heart Failure Center Accreditation Program (HF-CAP) is a hospital-level quality improvement intervention that includes standardized heart failure care processes, multidisciplinary team-based management, professional training, patient and caregiver education, structured discharge planning, post-discharge follow-up, and continuous performance monitoring and feedback.
  Arms: HF-CAP Intervention
Other: Usual Care — Usual care refers to the routine clinical management of patients hospitalized with heart failure according to local clinical practice and existing guidelines at each participating hospital. Hospitals assigned to this group do not implement the Heart Failure Center Accreditation Program (HF-CAP) or any additional structured quality improvement interventions beyond usual practice.
  Arms: Usual Care

SUMMARY:
Heart failure is a common and serious condition that affects millions of people in China and worldwide. Although effective treatments and clinical guidelines are available, the quality of heart failure care varies across hospitals, and many patients do not receive optimal management in real-world practice.

The Heart Failure Center Accreditation Program (HF-CAP) is a national quality improvement initiative in China designed to standardize and improve the diagnosis, treatment, and follow-up care of patients hospitalized with heart failure. This study aims to evaluate whether implementation of the HF-CAP program improves the quality of heart failure management and clinical outcomes compared with usual care.

This is a prospective, multicenter, cluster randomized controlled trial conducted in hospitals across China. Hospitals will be randomly assigned to either the HF-CAP intervention group or the usual care group. Adult patients hospitalized primarily for heart failure will be enrolled and followed for 12 months after discharge.

The main outcomes of this study are (1) a composite of heart failure rehospitalization or all-cause mortality within 12 months after discharge, and (2) a heart failure management quality score. Secondary outcomes include heart failure rehospitalization, all-cause rehospitalization, and all-cause mortality.

The results of this study are expected to provide high-quality evidence on whether hospital-based accreditation and quality improvement programs can improve the care and outcomes of patients with heart failure in real-world clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria for Participating Centers

* The participating center must be registered on the China Heart Failure Center website.Institutions applying for standard-level or primary-level heart failure center accreditation are required to have reported at least 300 or 100 heart failure cases, respectively, and must continuously report at least 10 or 8 heart failure cases per month, respectively.
* The participating center must have the capability to implement quality improvement measures.

Eligibility Criteria for Participants

* Age 18 years or older.
* Heart failure is the primary reason for hospitalization.

Whether hospitalization is due to heart failure will be determined by local investigators, but must meet the following criteria:

i. Presence of symptoms of heart failure (such as dyspnea or fatigue), signs of heart failure (such as elevated jugular venous pressure or peripheral edema), or laboratory or imaging evidence, including but not limited to: Pulmonary congestion on chest X-ray, Elevated natriuretic peptide levels, Echocardiographic evidence of structural or functional cardiac abnormalities. ii. Receipt of treatment targeting acute or chronic heart failure etiology, such as intravenous diuretics, vasodilators, positive inotropic agents, or coronary revascularization.

Exclusion Criteria:

* Presence of a life-threatening condition unrelated to heart failure with an expected life expectancy of less than 1 year (for example, advanced malignancy).
* Inability to complete the planned follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6240 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Composite of Heart Failure Rehospitalization or All-Cause Mortality | Within 12 months after hospital discharge
Heart Failure Management Quality Score | From baseline hospitalization to 12 months after discharge

SECONDARY OUTCOMES:
Time to First Heart Failure Rehospitalization | Within 12 months after hospital discharge
Number of Heart Failure Rehospitalizations | Within 12 months after hospital discharge
All-Cause Rehospitalization | Within 12 months after hospital discharge
All-Cause Mortality | Within 12 months after hospital discharge

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT07371780/Prot_SAP_ICF_000.pdf